CLINICAL TRIAL: NCT06737107
Title: Anatomical Segmentectomies for Early Stage Lung Cancer. A Multicenter Analysis of RATS, VATS and Open Approach
Brief Title: Multicenter Analysis of Different Approaches in Segmentectomies in Early-stage Lung Cancer
Acronym: ANASEGME
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: Istituto Clinico Humanitas (Other); Istituto Europeo di Oncologia (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pierluigi Novellis, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: 15/INT/2023
Record Dates: First submitted 2024-12-05; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Early Stage Lung Cancer (I and II); Non-Small Cell Lung Cancer
Keywords: Video-Assisted Thoracoscopic Surgery; open approach; Robot-Assisted Thoracoscopic Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group : Robotic Approach: Patients with a pre or post-operative diagnosis of NSCLC surgically treated with robotic segmentectomy from 1st January 2010 to the 31st to December 2023
- Control group: video-assisted thoracoscopic surgery (VATS) and open: Patients with a pre or post-operative diagnosis of NSCLC surgically treated with video-assisted thoracoscopic surgery (VATS) and open segmentectomy from 1st January 2010 to the 31st to December 2023

SUMMARY:
The study is a retrospective, observational and multicentric study. The study describes robotic segmentectomies performed in four referred centers, with the aim to assess the perioperative compilications of robotic segmentectomies compared to video-assisted thoracoscopic surgery (VATS) and open approach.

DETAILED DESCRIPTION:
Minimally invasive techniques have been gradually replacing open approach in the treatment of lung cancer. Video-assisted thoracoscopic surgery (VATS) was the first procedure to be developed in the thoracic field and is the most widespread. It has been associated with decreased postoperative pain, shorter recovery, decreased inflammatory response and improved tolerance to chemotherapy.

What is limiting video-assisted thoracoscopic surgery (VATS) spread is the steep learning curve, difficulties and discomfort to operate, suboptimal view and rigid instrumentation. These problems have been partially overcome by the Robotic technique (RATS).

This study aims to compare the perioperative complications of robotic segmentectomies to VATS and open approaches.

In addition, The secondary aim of the study is to analyze the duration of surgery, mediastinal and hilar lymph nodes dissection, rate of conversion of robotic approach compared to VATS, overall survival and disease free survival in the three different approaches.

The study is retrospective, observational and multicentric. The four centers involved are: IRCCS San Raffaele Hospital, IRCCS European Institute of Oncology - IEO, IRCCS Humanitas Research Hospital - ICH and the department of General Thoracic Surgery, Fondazione Policlinico Universitario "Agostino Gemelli" IRCCS, Università Cattolica del Sacro Cuore, Rome, Italy.

The population includes: all patients that underwent segmentectomies from the 1st January 2010 to the 31st of December 2023 treated with robotic segmentectomy and VATS or open segmentectomy, reaching a total of 472 cases of which 50 from our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Pre or post-operative diagnosis of NSCLC surgically treated with pulmonary segmentectomy from 1st January 2010 to the 31st to December 2023.
* Age > then 18 years at the moment of surgery

Exclusion Criteria:

* Age < then 18 years at the moment of surgery
* diagnosis other than NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent segmentectomies from the 1st January 2010 to the 31st of December 2023 treated with robotic segmentectomy (case) and video-assisted thoracoscopic (VATS) or open segmentectomy (control)
Sampling Method: Non-Probability Sample
Enrollment: 472 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The perioperative complications of robotic approach | from the surgery at 30-90 days after
  The investigators will measure the perioperative complications of robotic lung resection in patients with a pre or post-operative diagnosis of non-small cell lung cancer (NSCLC).
  Complications will be categorized according to the Clavien-Dindo scale.
The perioperative complication of video-assisted thoracoscopic surgery (VATS) approach | 30-90 days after surgery
  The investigators will measure the perioperative complications of video-assisted thoracoscopic surgery (VATS) appraoch in patients with a pre or post-operative diagnosis of non-small cell lung cancer (NSCLC).
  Complications will be categorized according to the Clavien-Dindo scale.
The perioperative complications of the open approach | 30-90 days after surgery
  The investigators will measure the perioperative complications of open approach in patients with a pre or post-operative diagnosis of non-small cell lung cancer (NSCLC). Complications will be categorized according to the Clavien-Dindo scale.

SECONDARY OUTCOMES:
Duration of surgery | up to 1 month
  Duration of the surgery based on the approach measured in minutes
Quality of lymphadenectomy | up to 1 month
  Number of lymphonodes station resected
Conversion rate | up to 1 month
  Number of surgery procedures converted
Survival analysis | up to 5 years
  Presence or absence of local and distant relapse

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Scientific Institute Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Policlinico Universitario Agostino Gemelli, Rome